CLINICAL TRIAL: NCT06161142
Title: The COHIR Study - a Non-interventional, Prospective, Single-center Investigation With Exploratory Data Analysis to Assess the Proportion of Patients With Hypophosphatasia Presenting at the Department of Rheumatology and Establishment of an Algorithm to HPP Diagnosis.
Brief Title: Characteristics of Hypophosphatasia in Adult Patients in Rheumatology
Acronym: COHIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, PD Dr. med. MuDr., University Hospital, Bonn
Other Study IDs: 407/21
Record Dates: First submitted 2023-07-03; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; Hypophosphatasemia; Musculoskeletal complaints; Rare disease; Genetic disorder; Alkaline phosphatase gene; ALP; ALP gene; Rheumatic disease; COHIR study; Prevalence; Diagnostic Algorithm; Metabolic bone diseases
MeSH Terms: conditions — Hypophosphatasia; Rare Diseases; Genetic Diseases, Inborn; Rheumatic Diseases; Bone Diseases, Metabolic | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persistant hypophosphatasemia: Patients with persistant hypophosphatasemia are highly suspicious for hypophosphatasia, and as such are the main focus of this study.
  In case of persistently low alkaline phosphatase (2nd measurement, 2-4 weeks after the 1st measurement) with normal serum calcium and phosphate values (exclusion of secondary hypophosphatemia due to e.g. rickets or malnutrition) and exclusion of other causes of secondary hypophosphatemia, genetic testing for a pathological ALP gene is performed as part of routine diagnostics.
  This study involves the structured recording of specific symptoms, the entire course of the disease since childhood, laboratory parameters and genetic testing.
  Interventions: Diagnostic Test: Second alkaline phosphatase measurement; Diagnostic Test: Extended laboratory diagnostics; Diagnostic Test: Symptom and clinical findings checklist for hypophosphatasia; Diagnostic Test: SF-36; Diagnostic Test: Short physical performance battery (SPPB) score; Diagnostic Test: Physical examination; Diagnostic Test: Recording of vital signs; Diagnostic Test: Bioelectrical Impedance Analysis; Diagnostic Test: Genetic testing of the alkaline phosphatase gene
- Transient hypophosphatasemia (Control group without hypophosphatasia): In patients, in which the initial hypophosphatasemia does not confirm with the second ALP testing, the former suspicion of hypophosphatasia must be discarded. With the exclusion of a hypophosphatasia (characterized by a persistant hypophosphatasemia among other criteria) this group of patients qualifies as a control group of patients without hypophosphatasia.
  Data from this control group will be analyzed in order to investigate patient historical, clinical and laboratory features that may help in the discrimination of hypophosphatasia patients against healthy individuals.
  Interventions: Diagnostic Test: Second alkaline phosphatase measurement; Diagnostic Test: Symptom and clinical findings checklist for hypophosphatasia; Diagnostic Test: SF-36; Diagnostic Test: Short physical performance battery (SPPB) score; Diagnostic Test: Physical examination; Diagnostic Test: Recording of vital signs; Diagnostic Test: Bioelectrical Impedance Analysis

INTERVENTIONS:
Diagnostic Test: Second alkaline phosphatase measurement — (2-4 weeks after the 1st measurement)
Diagnostic Test: Extended laboratory diagnostics — Laboratory testing investigating features that support the diagnosis of hypophosphatasia or exclude it by indicating secondary hypophosphatasemia for other reasons (including parameters such as serum calcium, inorganic serum phosphate, vitamin B6, vitamin B12, folic acid, bone-specific alkaline phosphatase, vitamin D3, and more).
  Groups: Persistant hypophosphatasemia
Diagnostic Test: Symptom and clinical findings checklist for hypophosphatasia — Checklist including numerous symptoms and clinical findings regarding the musculoskeletal system and non-musculoskeletal body parts
Diagnostic Test: SF-36 — Quality of life questionnaire
Diagnostic Test: Short physical performance battery (SPPB) score — The short physical performance battery is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older or disease-affected people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Diagnostic Test: Physical examination — A full rheumatological examination will be performed.
Diagnostic Test: Recording of vital signs — (including body temperature, blood pressure, heart rate)
Diagnostic Test: Bioelectrical Impedance Analysis — A body composition measurement by BIA (Bioelectrical Impedance Analysis [proportional mass of muscle, water and fat in kg]) will be performed.
Diagnostic Test: Genetic testing of the alkaline phosphatase gene — Investigation of mutations regarding the alkaline phosphatase gene
  Groups: Persistant hypophosphatasemia

SUMMARY:
With hypophosphatasia still being frequently overlooked and misdiagnosed, the primary aim of this prospective observational study is to determine the prevalence of hypophosphatasia in adult patients in rheumatology, and beyond that to establish an algorithm that promotes early hypophosphatasia detection in clinical practice.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a rare genetic disorder (1-3/300,000 severe cases in Europe) caused by one or more mutations in the alkaline phosphatase (ALP) gene. Hypomineralization results in symptoms such as arthralgias, insufficiency fractures, and poor dental status beginning in childhood. A fatal outcome is conceivable in circumstances of early infancy first presentation. In consistency with the musculoskeletal complaint pattern, HPP is far more common in the rheumatology patient population than in the general population.

However, HPP is still frequently misdiagnosed as some other form of bone disease (e.g., rickets, osteomalacia, or osteoporosis). Therefore, implementation of a clinically applicable algorithm for early hypophosphatasia detection is needed.

The primary aim of this prospective observational study is to determine the prevalence of hypophosphatasia in adult patients in rheumatology. Moreover, a further goal is to establish an algorithm that reliably separates adult HPP patients from other, rheumatologic and bone diseases.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Age > 18 years
* Clinical suspicion of hypophosphatasia
* Evidence of a pathological ALP value within the clinical routine screening

Exclusion Criteria:

* Failure to meet the inclusion criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient presenting at the University Hospital Bonn's rheumatology department with musculoskeletal complaints within the timeframe of the study conduct.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypophosphatasia in adult patients in rheumatology | 24 months
  The primary aim of this prospective observational study is to determine the prevalence of hypophosphatasia in adult patients presenting with musculoskeletal symptoms in rheumatology.

SECONDARY OUTCOMES:
Frequency of musculoskeletal pathology in hypophosphatasia patients in comparison with normal controls. | 24 months
  Frequency of musculoskeletal pathology in people with biochemistry suggestive of hypophosphatasia and positive ALP gene test as compared with normal controls.
Health-related quality of life: Short Form-36 | 24 months
  The possible score ranges from 0 to 100 points, where 0 points represent the greatest possible health limitation, while 100 points represent no health limitation at all.
Frequency of specific symptoms and clinical findings in patients with hypophosphatasia | 24 months
  This will be derived from the symptom and clinical findings checklist.
Frequency of specific patient history findings and the occurence of hypophosphatasia | 24 months
  Data will be derived from the medical history of hypophosphatasia patients (patient clinical data will be collected regarding the diagnosis, onset, progression, treatment course and outcome for patients with hypophosphatasia)
Correlation between physical performance abnormalities and hypophosphatasia | 24 months
  Physical performance is determined by standardized "short physical performance battery"
Correlation between body composition abnormalities and hypophosphatasia | 24 months
  Body composition is determined by bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin S. Schäfer, Dr. med., Principal Investigator — University Hospital of Bonn
Locations (1):
- Clinic of Internal Medicine III, Department of Oncology, Haematology, Rheumatology and Clinical Immunology, University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request